CLINICAL TRIAL: NCT02265094
Title: Associative Memory in ASD Without Mental Retardation : Study in EEG and Neuropsychology
Brief Title: Associative Memory in Autism Spectrum Disorder
Acronym: MEM-TA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Amiens University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2014- A00481-46
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Autistic Disorder
Keywords: Autism Spectrum Disorder; Development; Memory; ERD
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): Electroencephalography and neuropsychological tests in children with autism
  Interventions: Other: Electroencephalography; Behavioral: Neuropsychological assessment
- Control (Experimental): Electroencephalography and neuropsychological tests in children without autism
  Interventions: Other: Electroencephalography; Behavioral: Neuropsychological assessment

INTERVENTIONS:
Other: Electroencephalography — EEG recordings during memory tests
Behavioral: Neuropsychological assessment — patterns of eye gaze during cognitive tests

SUMMARY:
The aim of this study is to investigate the neural substrates of associative memory in Autism Spectrum Disorder using both behavioural and EEG assessments.

ELIGIBILITY:
Inclusion Criteria:

* Right handed children from 10 to 18 years old
* Informed consent signed by the legal representative and adolescent himself.
* Medical Examinations, psychopathology, and cognitive examination in accordance with inclusion and exclusion criteria specific to each population:

  * People with ASD:

    * Participants with ASD without mental retardation with a diagnosis in reference to the DSM V criteria
  * Controls : Participants without ASD

Main exclusion criteria:

* mental retardation,
* schizophrenia,
* ADHD,
* head injury with lost of consciousness

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-12-22 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Index of discrimination obtained with the task of associative memory | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc BALEYTE, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France